CLINICAL TRIAL: NCT04577118
Title: The iotaSOFT Insertion System Safety Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iotaMotion, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: iotaSOFT000001
Record Dates: First submitted 2020-09-22; First posted 2020-10-06 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-02

CONDITIONS: Cochlear Implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- iotaSOFT Insertion System (Other): The iotaSOFT Insertion System is a surgical device that aids the surgeon in implanting cochlear electrode arrays by controlling the speed and distance of implant insertion. All subjects enrolled in the trial will have the iotaSOFT Insertion System used during surgery.
  Interventions: Device: iotaSOFT Insertion System

INTERVENTIONS:
Device: iotaSOFT Insertion System — Enrolled subjects undergoing cochlear implant surgery will have the iotaSOFT Insertion System used by the surgeon to assist with implantation of the implant electrode array during the procedure.

SUMMARY:
Non-significant risk evaluation of the iotaSOFT Insertion System when used by a surgeon to assist with inserting a cochlear implant electrode array.

DETAILED DESCRIPTION:
This is a confirmatory study to assess successful peri-procedural use of the iotaSOFT Insertion System and potential adverse events that may be caused by use of the system during cochlear implant surgery.

ELIGIBILITY:
Key Inclusion Criteria:

* Candidate for cochlear implantation per indications
* Age 18 years or older

Key Exclusion Criteria:

* Prior cochlear implantation in ear to be treated
* Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode ray
* Craniofacial abnormality or abnormal cochlear/nerve anatomy on pre-operative CT or MR imaging
* Deafness due to lesions of the acoustic nerve or central auditory pathway
* Diagnosis of auditory neuropathy
* Active middle ear infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Gantz, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- iotaSOFT Insertion System: Purpose of this study is to evaluate safety of the iotaSOFT Insertion System when used by a surgeon to assist with inserting a cochlear implant array.
Period: Overall Study
Arm/Group | iotaSOFT Insertion System
Started | 25
Completed | 21
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Cochlear implant candidates 18 years and older at the time of surgery.
Groups:
- iotaSOFT Insertion System: Overall number of baseline participants: 25 Candidacy: Based on FDA indication for cochlear implantation Age: 18 years and older Language: English
Arm/Group | iotaSOFT Insertion System
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants] — 18 years and older Population: 4 subjects withdrawn
  Participants
    number analyzed (Participants) | 21
    <=18 years | 0
    Between 18 and 65 years | 15
    >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 4 subjects were withdrawn from the study.
  Participants
    number analyzed (Participants) | 21
    Female | 10
    Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants] — Population: 4 patients withdrawn
  Participants
    United States: number analyzed (Participants) | 21
    United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing a Peri-procedural Adverse Event Due to Use of the iotaSOFT Insertion System During Cochlear Implant Surgery
Description: Number of subjects experiencing a peri-procedural adverse event due to use of the iotaSOFT Insertion System and descriptions of reported adverse events. AEs will be summarized by type and number of subjects experiencing an event.
Time Frame: Day 0
Population: All enrolled subjects in study
Measure: Count of Participants; unit: Participants
Groups:
- iotaSOFT Insertion System: Overall number of baseline participants: 21 Candidacy: Based on FDA indication for cochlear implantation Age: 18 years and older Language: English
Arm/Group | iotaSOFT Insertion System
Number analyzed (Participants) | 21
Participants | 2

2. Secondary Outcome: Successful Surgical Use of the iotaSOFT Insertion System During Cochlear Implant Surgery as Measured by a Surgeon Utility Questionnaire. The Questionnaire Will be Used to Calculate the Proportion of Subjects in Which the Device Performed as Intended.
Description: The questionnaire will collect device handling data on proportion of subjects in which the device performed as intended, device utility, and ease of use.
Time Frame: Day 0
Population: All subjects enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | iotaSOFT Insertion System
Number analyzed (Participants) | 21
Participants | 21

3. Other Pre Specified Outcome: Procedural Duration of Time for Insertion of the Electrode Array (Mean, Range)
Description: The duration of time it takes for electrode array insertion will be measured
Time Frame: Day 0
Population: All enrolled and study completed subjects
Measure: Mean (Full Range); unit: Minutes
Arm/Group | iotaSOFT Insertion System
Number analyzed (Participants) | 21
Minutes | 2.5 [1.5 to 8]

4. Other Pre Specified Outcome: Proportion of Subjects in Which the Cochlear Implant Electrode Was in the Correct Position Post-procedure
Description: Post-procedural x-ray with cochlea view will be obtained to radiographically demonstrate positioning of the electrode.
Time Frame: Day 0
Population: Enrolled and completed subjects
Measure: Count of Participants; unit: Participants
Arm/Group | iotaSOFT Insertion System
Number analyzed (Participants) | 21
Participants | 21

5. Other Pre Specified Outcome: Adverse Events Reported During the Follow-up Period as Documented by Impedance and Neural Response Telemetry Testing. Adverse Events Will be Categorized by Type and Number of Participants Experiencing an Event.
Description: Potential risks and benefits of iotaSOFT will be assessed and characterized through data obtained during the post-surgical follow-up period while conducting impedance measurements and neural response telemetry.
Time Frame: 1 month
Population: Enrolled and completed subjects
Measure: Count of Participants; unit: Participants
Arm/Group | iotaSOFT Insertion System
Number analyzed (Participants) | 21
Participants | 0

ADVERSE EVENTS:
Time Frame: Surgery to 1 month post-operative
Description: Device related AEs and general AEs collected.
Arm/Group | iotaSOFT Insertion System
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 11/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iotaSOFT Insertion System (N=21)
Altered mental state (Psychiatric disorders) | 1 (1) — Altered mental state as reported by daughter to ER doctor. Patient has not returned for follow-up visit due to non-associated medical problems. Ongoing contact being made to clinic to reschedule.
Patient hospitalization following knee surgery (Surgical and medical procedures) | 1 (1) — Patient hospitalization following knee surgery. Knee pain pre-existing prior to surgery per patient/daughter report (ortho note history in medical file)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iotaSOFT Insertion System (N=21)
Resistance with iotaSOFT (Ear and labyrinth disorders) | 1 (1) — Resistance noted at 20mm with electrode array insertion attempted to 24mm. Intra-operative fluoroscopy showed electrode was coiled in the cochlea. After the tip fold over, per protocol, electrode was removed and inserted manually. Resolved.
No stimulation with device (Ear and labyrinth disorders) | 1 (1) — . Imaging was re-examined and identified a pre-existing temporal bone fracture crossing the internal auditory canal with scarring of the cochlear nerve (implant side). Subject withdrawn from study.
Drainage at implant site (Ear and labyrinth disorders) | 1 (1) — Patient reported drainage at implant site. This is identified risk of cochlear implantation surgery as captured in labeling and literature.
Bruising and dizziness (Ear and labyrinth disorders) | 1 (1) — Bruising and dizziness reported by patient following surgery. This is identified risk of cochlear implantation surgery as captured in labeling and literature.
CSF Leak (Ear and labyrinth disorders) | 1 (1) — Investigator used otologic drill for pilot hole for motor platform resulted in small CSF leak. Repaired and stopped with fascia and bone wax intraoperatively. No leak at closure. Surgery completed without further consequence or complications.
Dizziness (Ear and labyrinth disorders) | 1 (1) — No hospitalization necessary. Was seen by provider on 3-3-21. Recommended vestibular rehab locally. Based on time to onset of reported symptoms (74 days after surgery) it is unlikely this is related to use of the iotaSOFT during implantation.
Incision coming open at CI site as seen at 2-week post-op visit. (Ear and labyrinth disorders) | 1 (1) — Physician addressed by adding small additional suture. At subsequent visit (activation), healing issue resolved and activation occurred. This is identified risk of cochlear implantation surgery as captured in labeling and literature
Tinnitus (Ear and labyrinth disorders) | 1 (1) — Tinnitus when pushes on implant site. Patient reported tinnitus prior to surgery and by 1-month visit tinnitus 'better'. This is identified risk of cochlear implantation surgery as captured in labeling and literature.
Pain at incision (Ear and labyrinth disorders) | 1 (1) — Pain at incision w/ headache. This is identified risk of cochlear implantation surgery as captured in labeling and literature.
Swelling of face and eye area (Eye disorders) | 1 (1) — Swelling in face and eye area on side of implant site. This is identified risk of cochlear implantation surgery as captured in labeling and literature. Vastly improved at 2-week follow-up
Facial Stim (Ear and labyrinth disorders) | 1 (1) — Facial stim and poor electrode response. At follow-up appointment (activation) the facial stim resolved with widening the pulse width of signal. Electrodes 11 and 12 still no response as surgeon elected shallow insertion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT04577118/Prot_000.pdf